CLINICAL TRIAL: NCT06341829
Title: Assessment and Rehabilitation of Visuospatial and Affective Abilities in Parkinson Disease
Brief Title: Visuospatial and Affective Abilities in Parkinson Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Laura Culicetto, psychologist, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PRISM1
Record Dates: First submitted 2024-03-08; First posted 2024-04-02 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Parkinson Disease; Alexithymia; Visuospatial/Perceptual Abilities
MeSH Terms: conditions — Parkinson Disease; Affective Symptoms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Right prismatic adaptation (Experimental): This group will undergo right prismatic adaptation
  Interventions: Other: Prismatic adaptation
- Left prismatic adaptation (Experimental): This group will undergo left prismatic adaptation
  Interventions: Other: Prismatic adaptation
- Neutral prismatic adaptation (Sham Comparator): This group will undergo neutral lenses
  Interventions: Other: Prismatic adaptation

INTERVENTIONS:
Other: Prismatic adaptation — Participants will fit with prismatic goggles that deviate their visual field by 13° either leftward or rightward. They will seat in front of a white horizontal board on which three target dots (5 mm diameter) were positioned at 0, -10 and +10° from their body midline at a distance of 57 cm from their eyes. They will perform a total of 150 verbally instructed pointing movements with their right index finger towards the right (+10°) and left (-10°) targets in a pseudorandom order.

SUMMARY:
The aim of the study is to investigate whether prismatic adaptation (AP), a non-invasive neuromodulation technique, that involves the use of lenses that deviate the visual field, can modulate alexithyima and performance in visuospatial tasks in patients with Parkinson disease. Furthermore, brain activity during the prismatic adaptation and post-adaptation phases will be recorded using functional near-infrared spectroscopy (fNIRS) and high-density electroencephalography (HD-EEG).

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old;
* Right-handed;
* Diagnosis of idiopathic Parkinson's disease according to the UK Brain Bank criteria (Lyon and Pahwa, 2011);
* Hoehn and Yahr Stadium (Hoehn and Yahr, 1996) <2,5;
* Stable pharmacological treatment (dopaminergic therapy: dopamine agonists and Levo-dopa) in the last 6 weeks.

Exclusion Criteria:

* - Sensory-motor deficits that can hinder neuropsychological assessment;
* Visual system disorders (blindness, glaucoma);
* Atypical parkinsonisms;
* PD with dementia according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) (American Psychiatric Association).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-04-17 (Estimated); Primary Completion 2024-04-18 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Improve visuospatial skills; | 2 years
  Better performance in tests that evaluate visuospatial skills like line bisection test. The minimun value is 0 and the maximum is 3. Higher scores mean a worse outcome
Modulate alexithymia; | 2 years
  improvement in tests evaluating alexithymia such as TAS-20. The TAS 20 has scores that have a minimum of 20 and a maximum of 100. Scores greater than or equal to 61indicate high levels of alexithymia
Investigation of brain activity; | 2 years
  investigate the brain areas involved in the tasks with High Density Electroencephalography (EEG HD) and functional near infrared spectroscopy (fNIRS). The most active areas will be listed in a table

SECONDARY OUTCOMES:
Improve the quality of life with PDQ-39 questionnaire | 2 years
  Promote rewarding experiences that improve self-esteem, the perceived sense of self-efficacy, the quality of life measured with the Parkinson's disease questionnaire (PDQ-39).The minimum score is 0 which indicates the best quality of life A maximum score is 100 which indicates the worst quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Culicetto, Principal Investigator — IRCCS Centro Neurolesi Bonino Pulejo

IPD SHARING:
Plan to Share IPD: Undecided